CLINICAL TRIAL: NCT01534663
Title: Effects of Glutamine and Fish Oil on Muscle Function in Heart Failure (GlutFish-HF)
Brief Title: Supplementation of Glutamine and Fish Oil Versus Placebo in Patients With Heart Failure
Acronym: GLUTFISH-HF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Paolo Colombo, Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAE8356
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure
Keywords: Heart Failure; Skeletal Muscle Function; Metabolism; Inflammation; Glutamine; Fish oil; Muscle Function
MeSH Terms: conditions — Heart Failure; Inflammation | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo for fish oil will be safflower oil. For glutamine, soy powder will serve as the placebo.
  Interventions: Drug: Placebo
- Glutamine/Fishoil (Active Comparator): 3.285 g of EPA and 3.285 g of Docosahexaenoic acid (DHA) and L-alanyl-glutamine (8g/d).
  Interventions: Drug: Glutamine and Fish Oil Supplementation

INTERVENTIONS:
Drug: Glutamine and Fish Oil Supplementation — This is a prospective, randomized double-blind, placebo-controlled study design. 38 subjects will be randomized to two groups (19 patients in each group), one taking active fish oil and glutamine supplementation and the other taking placebo for 90 days.
  Arms: Glutamine/Fishoil
Drug: Placebo — This is a prospective, randomized double-blind, placebo-controlled study design. 38 subjects will be randomized to two groups (19 patients in each group), one taking active fish oil and glutamine supplementation and the other taking placebo for 90 days.
  Arms: Placebo

SUMMARY:
The aim of this study is to determine whether supplementation of glutamine and fish oil can improve peripheral skeletal muscle function and metabolism in patients with heart failure. The investigators propose a randomized, double-blind, placebo controlled study comparing the combined supplementation of fish oil and glutamine with placebo in patients with stable heart failure. 30 patients with heart failure will be randomized to either receiving 6.5 g fish oil/d and 8 g glutamine/d (n=15) or placebo (n=15) for 90 days. The primary outcome in this study is the change in muscle functional capacity measured as changes in maximum muscle strength and fatigability, peak VO2 and exercise time after supplementation. A secondary outcome is the measurement of systemic and local markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years,
* left ventricular ejection fraction less than or equal to 35%,
* stable on standard HF medications, and
* optimal medical therapy.

Exclusion Criteria:

* major cardiovascular events,
* procedures in the last 6 months,
* dementia,
* presence of cardiovascular diseases that may lead to harm if the patient took part in the study (congenital heart disease, long QT syndrome, hypertrophic cardiomyopathy, active myocarditis).

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo C. Colombo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Shahzad K, Chokshi A, Schulze PC. Supplementation of glutamine and omega-3 polyunsaturated fatty acids as a novel therapeutic intervention targeting metabolic dysfunction and exercise intolerance in patients with heart failure. Curr Clin Pharmacol. 2011 Nov;6(4):288-94. doi: 10.2174/157488411798375958. PMID 22082326
- [Derived] Wu C, Kato TS, Ji R, Zizola C, Brunjes DL, Deng Y, Akashi H, Armstrong HF, Kennel PJ, Thomas T, Forman DE, Hall J, Chokshi A, Bartels MN, Mancini D, Seres D, Schulze PC. Supplementation of l-Alanyl-l-Glutamine and Fish Oil Improves Body Composition and Quality of Life in Patients With Chronic Heart Failure. Circ Heart Fail. 2015 Nov;8(6):1077-87. doi: 10.1161/CIRCHEARTFAILURE.115.002073. Epub 2015 Aug 12. PMID 26269566

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventeen participants were randomized to the active treatment group and 14 to the placebo group. Three participants dropped out in the active treatment group. Two participants dropped out of the placebo group. A total of 14 participants completed the trial in the active treatment group and 12 in the placebo group.
Groups:
- Glutamine/Fishoil: 3.285 g of EPA and 3.285 g of DHA and L-alanyl-glutamine (8g/d).
  Glutamine and Fish Oil Supplementation: This is a prospective, randomized double-blind, placebo-controlled study design. 38 subjects will be randomized to two groups (19 patients in each group), one taking active fish oil and glutamine supplementation and the other taking placebo for 90 days.
Period: Overall Study
Arm/Group | Placebo | Glutamine/Fishoil
Started | 14 | 17
Completed | 12 | 14
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Glutamine/Fishoil | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (2) | 59 (3) | 59 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 9 | 12 | 21
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Baseline Skeletal Muscle Function Capacity- Isometric Contractions (PKTQ/BW)
Description: For isometric contractions, participants contracted against a constant 60-degree angle at the knee (dominant leg) and a constant 30 degree angle at the elbow (dominant arm) for 6 seconds. Participants alternated between flexion and extension, 3 repetitions each with a 30 second rest period between each. Data was collected to determine peak torque to body weight (peak torque (PKTQ)/ body weight (BW)).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Percent
  Knee: Extension | 177 (18) | 196 (10)
  Knee: Flexion | 76 (6) | 90 (5)
  Elbow: Extension | 65 (6) | 59 (4)
  Elbow: Flexion | 74 (7) | 71 (4)

2. Primary Outcome: 90 Day Skeletal Muscle Function Capacity- Isometric Contractions (PKTQ/BW)
Description: as for outcome 1
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Percent
  Knee: Extension | 200 (20) | 206 (11)
  Knee: Flexion | 90 (8) | 90 (5)
  Elbow: Extension | 64 (6) | 61 (4)
  Elbow: Flexion | 74 (6) | 74 (4)

3. Primary Outcome: Baseline Muscle Function Capacity- Isokinetic Contractions (PKTQ/BW)
Description: For isokinetic contractions, subjects performed flexion and extension movements at the knee and elbow for 5 repetitions at a speed of 60 degrees/second. This was followed by a rest period of 2.5 minutes. For the second isokinetic protocol, subjects performed 25 repetitions of flexion and extension movements at the knee and elbow at a speed of 180 degrees/second.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Percent
  Knee: Extension, 5 repetitions | 147 (17) | 153 (8)
  Knee: Flexion, 5 repetitions | 61 (6) | 70 (5)
  Elbow: Extension, 5 repetitions | 46 (5) | 42 (3)
  Elbow: Flexion, 5 repetitions | 61 (6) | 54 (3)
  Knee: Extension, 25 repetitions | 103 (10) | 105 (7)
  Knee: Flexion, 25 repetitions | 55 (5) | 96 (33)
  Elbow: Extension, 25 repetitions | 37 (3) | 35 (2)
  Elbow: Flexion, 25 repetitions | 56 (5) | 50 (3)

4. Primary Outcome: 90 Day Muscle Function Capacity- Isokinetic Contractions (PKTQ/BW)
Description: as for outcome 3
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Percent
  Knee: Extension, 5 repetitions | 173 (20) | 160 (9)
  Knee: Flexion, 5 repetitions | 76 (9) | 77 (4)
  Elbow: Extension, 5 repetitions | 48 (5) | 46 (2)
  Elbow: Flexion, 5 repetitions | 56 (4) | 57 (3)
  Knee: Extension, 25 repetitions | 115 (10) | 108 (6)
  Knee: Flexion, 25 repetitions | 58 (4) | 67 (3)
  Elbow: Extension, 25 repetitions | 38 (4) | 36 (2)
  Elbow: Flexion, 25 repetitions | 55 (4) | 51 (3)

5. Primary Outcome: Baseline Muscle Function Capacity- Isokinetic Contractions (Work (WK)/Body Weight (BW))
Description: as for outcome 3
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Percent
  Knee: Extension, 5 repetitions | 132 (15) | 137 (8)
  Knee: Flexion, 5 repetitions | 61 (9) | 70 (6)
  Elbow: Extension, 5 repetitions | 51 (6) | 47 (4)
  Elbow: Flexion, 5 repetitions | 70 (7) | 65 (4)
  Knee: Extension, 25 repetitions | 100 (11) | 102 (7)
  Knee: Flexion, 25 repetitions | 41 (6) | 46 (6)
  Elbow: Extension, 25 repetitions | 38 (4) | 36 (3)
  Elbow: Flexion, 25 repetitions | 63 (6) | 55 (3)

6. Primary Outcome: 90 Days Muscle Function Capacity- Isokinetic Contractions (Work (WK)/Body Weight (BW))
Description: as for outcome 3
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Percent
  Knee: Extension, 5 repetitions | 157 (17) | 149 (9)
  Knee: Flexion, 5 repetitions | 78 (12) | 80 (5)
  Elbow: Extension, 5 repetitions | 54 (6) | 54 (3)
  Elbow: Flexion, 5 repetitions | 68 (5) | 71 (4)
  Knee: Extension, 25 repetitions | 111 (11) | 108 (7)
  Knee: Flexion, 25 repetitions | 51 (6) | 55 (4)
  Elbow: Extension, 25 repetitions | 41 (4) | 39 (2)
  Elbow: Flexion, 25 repetitions | 60 (5) | 58 (3)

7. Primary Outcome: Baseline Muscle Function Capacity- Isokinetic Contractions (Total Work)
Description: as for outcome 3
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Joules
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Joules
  Knee: Extension, 5 repetitions | 477 (64) | 537 (50)
  Knee: Flexion, 5 repetitions | 209 (35) | 264 (36)
  Elbow: Extension, 5 repetitions | 189 (23) | 184 (19)
  Elbow: Flexion, 5 repetitions | 280 (35) | 261 (22)
  Knee: Extension, 25 repetitions | 1551 (200) | 1776 (185)
  Knee: Flexion, 25 repetitions | 552 (102) | 742 (118)
  Elbow: Extension, 25 repetitions | 590 (72) | 612 (65)
  Elbow: Flexion, 25 repetitions | 1108 (141) | 992 (74)

8. Primary Outcome: 90 Day Muscle Function Capacity- Isokinetic Contractions (Total Work)
Description: as for outcome 3
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: Joules
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Joules
  Knee: Extension, 5 repetitions | 586 (69) | 603 (51)
  Knee: Flexion, 5 repetitions | 277 (44) | 319 (33)
  Elbow: Extension, 5 repetitions | 209 (26) | 193 (18)
  Elbow: Flexion, 5 repetitions | 272 (27) | 283 (15)
  Knee: Extension, 25 repetitions | 1806 (176) | 1816 (168)
  Knee: Flexion, 25 repetitions | 765 (99) | 813 (99)
  Elbow: Extension, 25 repetitions | 655 (83) | 598 (50)
  Elbow: Flexion, 25 repetitions | 1079 (118) | 987 (55)

9. Primary Outcome: Baseline Muscle Function Capacity- Isokinetic Contractions (Average Power)
Description: as for outcome 3
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Watts
  Knee: Extension, 5 repetitions | 65 (10) | 75 (33)
  Knee: Flexion, 5 repetitions | 26 (5) | 33 (5)
  Elbow: Extension, 5 repetitions | 24 (3) | 23 (3)
  Elbow: Flexion, 5 repetitions | 35 (4) | 32 (3)
  Knee: Extension, 25 repetitions | 106 (14) | 121 (13)
  Knee: Flexion, 25 repetitions | 26 (7) | 46 (7)
  Elbow: Extension, 25 repetitions | 37 (5) | 38 (5)
  Elbow: Flexion, 25 repetitions | 64 (9) | 57 (5)

10. Primary Outcome: 90 Day Muscle Function Capacity- Isokinetic Contractions (Average Power)
Description: as for outcome 3
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Watts
  Knee: Extension, 5 repetitions | 80 (9) | 84 (7)
  Knee: Flexion, 5 repetitions | 37 (6) | 41 (5)
  Elbow: Extension, 5 repetitions | 26 (3) | 25 (2)
  Elbow: Flexion, 5 repetitions | 34 (4) | 34 (2)
  Knee: Extension, 25 repetitions | 128 (13) | 140 (15)
  Knee: Flexion, 25 repetitions | 50 (7) | 56 (7)
  Elbow: Extension, 25 repetitions | 40 (6) | 36 (4)
  Elbow: Flexion, 25 repetitions | 62 (8) | 57 (4)

11. Primary Outcome: Baseline Muscle Function Capacity- Isokinetic Contractions (Time to Peak Torque)
Description: as for outcome 3
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
msec
  Knee: Extension, 5 repetitions | 526 (44) | 494 (27)
  Knee: Flexion, 5 repetitions | 828 (104) | 945 (84)
  Elbow: Extension, 5 repetitions | 426 (50) | 344 (26)
  Elbow: Flexion, 5 repetitions | 806 (89) | 1003 (76)
  Knee: Extension, 25 repetitions | 195 (12) | 212 (27)
  Knee: Flexion, 25 repetitions | 399 (61) | 546 (11)
  Elbow: Extension, 25 repetitions | 376 (58) | 417 (50)
  Elbow: Flexion, 25 repetitions | 435 (52) | 426 (42)

12. Primary Outcome: 90 Day Muscle Function Capacity- Isokinetic Contractions (Time to Peak Torque)
Description: as for outcome 3
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
msec
  Knee: Extension, 5 repetitions | 404 (37) | 456 (27)
  Knee: Flexion, 5 repetitions | 729 (45) | 780 (93)
  Elbow: Extension, 5 repetitions | 429 (65) | 469 (45)
  Elbow: Flexion, 5 repetitions | 808 (77) | 996 (80)
  Knee: Extension, 25 repetitions | 186 (12) | 177 (12)
  Knee: Flexion, 25 repetitions | 366 (53) | 507 (32)
  Elbow: Extension, 25 repetitions | 417 (54) | 314 (47)
  Elbow: Flexion, 25 repetitions | 420 (48) | 426 (43)

13. Primary Outcome: Percent Change in Peak Effort Oxygen Consumption
Description: Peak effort oxygen consumption (VO2 max) is measured using Cardiopulmonary Exercise Testing (CPET).
Time Frame: Baseline to 90 Days
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
Percent | 7.9 (4.7) | 0.1 (0.7)

14. Secondary Outcome: Baseline Systemic and Local Inflammation
Description: Systemic and local marker of inflammation as measured by tumor necrosis factor-alpha, units pg/mL
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
pg/mL | 3.4 (0.6) | 3.1 (0.8)

15. Secondary Outcome: 90 Day Systemic and Local Inflammation
Description: Systemic and local marker of inflammation as measured by tumor necrosis factor-alpha, units pg/mL
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Glutamine/Fishoil
Number analyzed (Participants) | 12 | 14
pg/mL | 2.5 (0.4) | 3.3 (0.5)

ADVERSE EVENTS:
Time Frame: 90 Days
Arm/Group | Placebo | Glutamine/Fishoil
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 2/12 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Glutamine/Fishoil (N=14)
Diarrhea (Gastrointestinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes